CLINICAL TRIAL: NCT06399302
Title: Prospective Multicenter Research on Donor and Recipient Management Strategies to Improve Lung Transplant Outcomes: PROMISE-Lung Study
Brief Title: Prospective Multicenter Research on Donor and Recipient Management Strategies to Improve Lung Transplant Outcomes
Acronym: PROMISE
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00114566; U24HL163122 (NIH); PROMISE Study (Other: LTC-DCC)
Record Dates: First submitted 2024-05-01; First posted 2024-05-03 (Actual); Last update posted 2025-07-07 (Actual); Status verified 2025-07

CONDITIONS: Lung Transplant; Complications; Lung Transplant; Infection or Inflammation; Lung Transplant Rejection; Lung Transplant Failure
MeSH Terms: conditions — Infections; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The DCC will establish the centralized biorepository for the PROMISE-Lung Study at the University of Pennsylvania (Penn). Each specimen will be labeled with the study, sample ID, time-point, specimen type, and a unique barcode ID. Following local site processing, specimens will be locally stored at -80ᵒC at the participating site. Samples will then be batched and shipped on dry ice overnight to Penn at regular intervals. Shipments will be tracked to ensure arrival in a timely manner. Once received at Penn, all biological specimens for the cohort will be scanned into the laboratory information management system (LIMs) and stored at -80ᵒC. Biospecimens sent to Penn will be stored for future research studies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lung transplant donors and recipients: Lung transplant donors and adult (18 years and up) lung transplant candidates and recipients

SUMMARY:
This project aims to collect detailed clinical data, blood samples, and patient-reported outcomes from 2,600 lung transplant candidates, donors, and recipients at Lung Transplant Centers. The goal is to create a robust resource for various research objectives, including studying the impact of variations in donor and medical practices on clinical outcomes. The project also seeks to identify serum biomarkers associated with or predictive of specific post-transplant complications and conditions.

DETAILED DESCRIPTION:
This is an observational, prospective, multicenter cohort study of 2,600 lung transplant donors and adult (18 years and older) lung transplant candidates and recipients that will collect longitudinal clinical data, and serial biological (blood) specimens and PROs to support a broad range of clinical and translational future research. Data and biospecimens will be rigorously collected and monitored to ensure high quality future studies that will address unmet needs and optimal management at each stage of the transplant journey from listing, to donor selection, to postoperative management. Subjects are recruited to the study either prior to undergoing lung transplant at the time of listing or within 30 days of having undergone a lung transplant at one of the enrolling centers.

The study design will generally follow the SOC practices at each center to minimize additional research related visits. Participants will follow the SOC transplant protocols at each site. Every attempt will be made by the site to collect study data and research specimens from participants at the time of SOC visits. Participation in this study will include scheduled data extraction or data transfers at specified time intervals, serial prospective blood collection (including plasma, serum), recipient DNA sample collection (with donor DNA sample collection optional), and PRO measures.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and provide informed consent
2. ≥ 18 years of age at the time of written informed consent
3. Anticipated listing or listed for a single or bilateral cadaveric donor lung transplant or having received a lung transplant within 30 days

   * Participants undergoing repeat lung transplantation or multi-organ transplantation are eligible if they meet the inclusion/exclusion criteria.

Exclusion Criteria:

1. Unwillingness of a participant or legally authorized representative (LAR) to give written informed consent or comply with study protocol
2. Pregnancy or plans to become pregnant
3. Past or current medical problems or findings from physical examination or laboratory testing, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung transplant donors and adult (18 years and up) lung transplant candidates and recipients
Sampling Method: Non-Probability Sample
Enrollment: 2600 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants enrolled and critical variable completeness | 3 years
  To collect detailed clinical data, blood samples (including DNA), and PROs in 2,600 lung transplant candidates, donors, and recipients across the participating LTC centers to create a robust resource that will support a broad range of additional future clinical and translational research objectives
Number of PROs collected per patient | 3 years
  To collect clinical data and PROs that will specifically support future research studies to determine how variation in donor, surgical, or medical management practices across the participating LTC centers are associated with specific differences in relevant clinical outcomes such as PGD, AR, AMR, ALAD, post-transplant infections, PROs including health-related quality of life, or one-year survival.
Number of specimens per participant collected | 3 years
  To collect clinical data and biosamples that will specifically support future research studies to identify serum biomarkers that are associated with or predict the development of PGD, AR, AMR, ALAD, or CLAD.

CONTACTS AND LOCATIONS:
Overall Officials: Scott M Palmer, MD, MHS, Principal Investigator — Duke University School of Medicine, Department of Medicine; Jason D Christie, MD, MSCE, Principal Investigator — University of Pennsylvania; Megan L Neely, PhD, Principal Investigator — Duke University School of Medicine, Department of Biostatistics and Bioinformatics
Locations (17):
- United States (16):
  - University of California Los Angeles, Los Angeles, California
  - University of California at San Francisco, San Francisco, California
  - University of Miami, Miami, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Womens Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - New York University, New York, New York
  - Columbia University, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Inova Fairfax Hospital, Falls Church, Virginia
  - University of Washington, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- University Health Network, Toronto, Canada

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed, information about the study, including study data, will be submitted to the NIH data repository. NHLBI's BioData Catalyst will be used for data, and BioLINCC will be used for biosample deposition after study completion.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data from each cycle of an examination or follow-up component are prepared by the DCC and sent to the NHLBI Program Officer for distribution no later than 3 years after the completion of each examination or follow-up cycle or 2 years after the baseline, follow-up, genetic, ancillary study, or other data set is finalized within the study for analysis for use in publication, whichever comes first.
Access Criteria: The overall governance of the protocol is under the guidance of the NHLBI and the steering committee, composed of members of the DCC and UO1 site representatives. Future studies using these sample will be governed by an ancillary committee of the steering committee.
  In addition, further analysis using this data may occur via ancillary studies that are submitted separately for IRB review.
  https://biodatacatalyst.nhlbi.nih.gov/ https://biolincc.nhlbi.nih.gov/home/